CLINICAL TRIAL: NCT05447689
Title: Integrative-Mind-Body Skills Group for Mood Management Among Medical Graduate Students
Brief Title: Mind-Body Skills Group for Graduate Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-02024481
Record Dates: First submitted 2022-06-29; First posted 2022-07-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Mood Change; Depressive Symptoms; Anxiety Generalized
Keywords: Mind-Body Skills Group Intervention; Graduate student mental health; Medical student mental health
MeSH Terms: conditions — Depression; Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: The intervention will be delivered across eight weeks (1 session weekly).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrative-Mind-Body Skills Group (Experimental): Treatment group
  Interventions: Behavioral: Integrative-Mind-Body Skills Group
- Control (No Intervention): Control group: Treatment-As-Usual (TAU) and mind-body skills reading materials.

INTERVENTIONS:
Behavioral: Integrative-Mind-Body Skills Group — Integrative-Mind-Body Skills Group (I-MBS-G) is an 8-week group that teaches skills to build inner resources for effective mood management. This group incorporates a holistic approach to wellness through meditation and mindfulness practices, guided imagery, breath and body awareness, relaxation techniques, self-reflection, and mindfulness-based cognitive-behavioral skills. Mind-body approaches have demonstrated effectiveness in reducing stress mood symptoms and improving quality of life.
  Arms: Integrative-Mind-Body Skills Group

SUMMARY:
Integrative-Mind-Body Skills Group (I-MBS-G) is an 8-week group that teaches skills to build inner resources for effective mood management. This group incorporates a holistic approach to wellness through meditation and mindfulness practices, guided imagery, breath and body awareness, and relaxation techniques. Mind-body approaches have demonstrated effectiveness in reducing stress mood symptoms and improving quality of life. The study hypothesis is that the Mind-Body Skills taught in the group will reduce mood symptoms in graduate and medical students.

DETAILED DESCRIPTION:
Study Design: This study will identify medical graduate students interested in participating in an Integrative-Mind-Body Skills Group (I-MBS-G) to strengthen inner resources to effectively navigate complex and stressful daily events to promote mental and physical health and well-being. This study is a pilot randomized controlled trial; participants will be randomized to the intervention or control group. The control group will receive Treatment-As-Usual (TAU) and mind-body skills reading materials.

Primary Objective: Assess the feasibility and acceptability of an I-MBS-G intervention for medical graduate students using the MBSG Feedback Program Questionnaire.

Secondary Objectives: Assess preliminary effectiveness of I-MBS-G on anxiety symptoms (i.e., improvements on anxiety symptoms)

Exploratory Objectives: Assess preliminary effectiveness of I-MBS-G on depression symptoms (i.e., improvements on depression symptoms)

ELIGIBILITY:
Inclusion Criteria:

* Students screened and admitted to the Student Mental Health Program.
* Age 18 or older
* A score of ≥ 4 on the Generalized Anxiety Disorder scale (GAD-7)
* Able to attend weekly meeting times

Exclusion Criteria:

* Active SI
* Current mania
* Active psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The Integrative-Mind-Body Skills Group program evaluation measures the acceptability of the Integrative-Mind-Body Skills Group Program. | Week 9
  The Integrative-Mind-Body Skills Group program evaluation is a quantitative self-report survey assessing the acceptability of the Integrative-Mind-Body Skills Group measured at Week 9. The Integrative-Mind-Body Skills Group evaluation uses three items measured on a 5-point Likert scale and one item measured on a 3-point Likert scale. Score range: 4- 18; acceptability = a sum score of 14 or greater; unacceptability = a sum score of 4.
The Integrative-Mind-Body Skills Group program evaluation measures the feasibility of the Integrative-Mind-Body Skills Group Program. | Week 9
  The Integrative-Mind-Body Skills Group program evaluation is a quantitative self-report survey assessing the feasibility of the Integrative-Mind-Body Skills Group measured at Week 9. To evaluate the feasibility of the Integrative-Mind-Body Skills Group, the number of sessions attended is measured by one item. There are eight sessions in the program. Score range: 1- 8; feasibility = score of 5 sessions or greater.

SECONDARY OUTCOMES:
Change from Baseline (week 0) in Anxiety symptoms as measured in the Generalized Anxiety Disorder (GAD-7) at Weeks 9 and 13. | Week 0, Week 9 and Week 13
  The Generalized Anxiety Disorder scale is a validated, self-report instrument assessing the severity of anxiety symptoms across the previous two weeks. Score range: 0-21; minimal anxiety 0-4; mild anxiety 5-9; moderate 10-14; Moderately severe depression 15-10; Severe anxiety - a score greater than 15. Change = (Week 13 score - Week 0 score). Change = (Week 9 score - Week 0 score).

OTHER OUTCOMES:
Change from Baseline (week 0) in Depressive symptoms as measured on the Patient Health Questionnaire (PHQ-9) at Weeks 9 and 13. | Week 0, Week 9 and Week 13
  The Patient Health Questionnaire (PHQ-9) is a validated, self-report instrument assessing the severity of depressive symptoms across the previous two weeks. Score range: 0-27; minimal depression 0-4; mild depression 5-9; moderate depression 10-14; Moderately severe depression 15-10; Severe depression 20-27. Change = (Week 13 score - Week 0 score). Change = (Week 9 score - Week 0 score).

CONTACTS AND LOCATIONS:
Overall Officials: Suza C Scalora, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christophers B, Nieblas-Bedolla E, Gordon-Elliott JS, Kang Y, Holcomb K, Frey MK. Mental Health of US Medical Students During the COVID-19 Pandemic. J Gen Intern Med. 2021 Oct;36(10):3295-3297. doi: 10.1007/s11606-021-07059-y. Epub 2021 Aug 5. No abstract available. PMID 34355345
- [Background] Mousa OY, Dhamoon MS, Lander S, Dhamoon AS. The MD Blues: Under-Recognized Depression and Anxiety in Medical Trainees. PLoS One. 2016 Jun 10;11(6):e0156554. doi: 10.1371/journal.pone.0156554. eCollection 2016. PMID 27286249
- [Background] Rotenstein LS, Ramos MA, Torre M, Segal JB, Peluso MJ, Guille C, Sen S, Mata DA. Prevalence of Depression, Depressive Symptoms, and Suicidal Ideation Among Medical Students: A Systematic Review and Meta-Analysis. JAMA. 2016 Dec 6;316(21):2214-2236. doi: 10.1001/jama.2016.17324. PMID 27923088
- [Background] Compton MT, Carrera J, Frank E. Stress and depressive symptoms/dysphoria among US medical students: results from a large, nationally representative survey. J Nerv Ment Dis. 2008 Dec;196(12):891-7. doi: 10.1097/NMD.0b013e3181924d03. PMID 19077856
- [Background] Goebert D, Thompson D, Takeshita J, Beach C, Bryson P, Ephgrave K, Kent A, Kunkel M, Schechter J, Tate J. Depressive symptoms in medical students and residents: a multischool study. Acad Med. 2009 Feb;84(2):236-41. doi: 10.1097/ACM.0b013e31819391bb. PMID 19174678
- [Background] Dyrbye LN, Thomas MR, Huschka MM, Lawson KL, Novotny PJ, Sloan JA, Shanafelt TD. A multicenter study of burnout, depression, and quality of life in minority and nonminority US medical students. Mayo Clin Proc. 2006 Nov;81(11):1435-42. doi: 10.4065/81.11.1435. PMID 17120398
- [Background] Dyrbye LN, Thomas MR, Huntington JL, Lawson KL, Novotny PJ, Sloan JA, Shanafelt TD. Personal life events and medical student burnout: a multicenter study. Acad Med. 2006 Apr;81(4):374-84. doi: 10.1097/00001888-200604000-00010. PMID 16565189
- [Background] Dyrbye LN, Thomas MR, Massie FS, Power DV, Eacker A, Harper W, Durning S, Moutier C, Szydlo DW, Novotny PJ, Sloan JA, Shanafelt TD. Burnout and suicidal ideation among U.S. medical students. Ann Intern Med. 2008 Sep 2;149(5):334-41. doi: 10.7326/0003-4819-149-5-200809020-00008. PMID 18765703
- [Background] Dahlin M, Joneborg N, Runeson B. Performance-based self-esteem and burnout in a cross-sectional study of medical students. Med Teach. 2007 Feb;29(1):43-8. doi: 10.1080/01421590601175309. PMID 17538833
- [Background] Gordon JS. Mind-body skills groups for medical students: reducing stress, enhancing commitment, and promoting patient-centered care. BMC Med Educ. 2014 Sep 22;14:198. doi: 10.1186/1472-6920-14-198. PMID 25245341
- [Background] Ayala EE, Winseman JS, Johnsen RD, Mason HRC. U.S. medical students who engage in self-care report less stress and higher quality of life. BMC Med Educ. 2018 Aug 6;18(1):189. doi: 10.1186/s12909-018-1296-x. PMID 30081886
- [Background] Yonker JE, Schnabelrauch CA, Dehaan LG. The relationship between spirituality and religiosity on psychological outcomes in adolescents and emerging adults: a meta-analytic review. J Adolesc. 2012 Apr;35(2):299-314. doi: 10.1016/j.adolescence.2011.08.010. Epub 2011 Sep 14. PMID 21920596
- [Background] Yotter, C. N., & Swank, M. (2017). The impact of spirituality and stress on the health of emerging adults. SUURJ: Seattle University Undergraduate Research Journal, 1(1), 17.
- [Background] Liu, C., Beauchemin, J., Wang, X., & Lee, M. Y. (2018). Integrative body-mind-spirit (I-BMS) interventions for posttraumatic stress disorder (PTSD): A review of the outcome literature. Journal of Social Service Research, 44(4), 482-493.
- [Background] King AP, Erickson TM, Giardino ND, Favorite T, Rauch SA, Robinson E, Kulkarni M, Liberzon I. A pilot study of group mindfulness-based cognitive therapy (MBCT) for combat veterans with posttraumatic stress disorder (PTSD). Depress Anxiety. 2013 Jul;30(7):638-45. doi: 10.1002/da.22104. Epub 2013 Apr 17. PMID 23596092